CLINICAL TRIAL: NCT05727774
Title: Effect of Hot Versus Neutral Water for Heat Acclimatation and Sport Performance During a Water Biking Training Protocol : Controlled Randomised Study
Brief Title: Effect of Water Biking in Hot Versus Neutral Water for Heat Acclimatation
Acronym: THERMIDOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL22_0076
Record Dates: First submitted 2023-01-12; First posted 2023-02-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: Healthy; Heat Exposure
Keywords: Water biking; Acclimatization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot water condition (Experimental): Participants do the water biking training for two weeks, 1 hour a day, in hot water temperature (35°C)
  Interventions: Other: Water Biking in hot water condition
- Neutral water condition (Sham Comparator): Participants do the water biking training for two weeks, 1 hour a day, in neutral water temperature (25°C)
  Interventions: Other: Water Biking in neutral water condition

INTERVENTIONS:
Other: Water Biking in hot water condition — Training protocol includes 10 water biking sessions in hot water temperature (35°C) for this group
  Arms: Hot water condition
Other: Water Biking in neutral water condition — Training protocol includes 10 water biking sessions in neutral water temperature (25°C) for this group
  Arms: Neutral water condition

SUMMARY:
The goal of this clinical trial is to compare the efficiency of water biking training in hot (35°C) versus neutral (25°C) temperature water to elicite heat acclimation in healthy recreative athletes.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the efficiency of water biking training in hot (35°C) versus neutral (25°C) temperature water to elicite heat acclimation in healthy recreative athletes. The main questions it aims to answer are:

* Does the water biking training protocol in hot versus neutral temperature water improve the time trial in an artificially hot and humid indoor environment?
* Does the water biking training protocol in hot versus neutral temperature water improve the VO2 max performance and force/velocity profile in neutral indoor environment?
* What are the main acclimation adaptations (central and cutaneous temperature), heart rate, cardiac function, sweating quality, sleep quality, haematologic profile.

Participants will have to do pre and post training tests in both normal environment (cardiorespiratory stress test, force/velocity profile test, echocardiography) and artificially hot and humid indoor environment (time trial). The training protocols consists in 10 sessions of 1 hour of water bike aerobic training (5 times a week for 2 weeks) at an intensity based on the heart rate corresponding to the 1st respiratory threshold, in hot (interventional group IG: 35°C) versus neutral (control group CG: 25°C) water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people
* Sports practicing

Exclusion Criteria:

* Acclimatation already done (recent training in hot and/or humid) less than 2 months
* Heart disease recent or non controlled
* Heat intolerance
* Water phobia or inable to swim

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Change of the distance traveled (meter) on a Time Trial between pre and post training tests in hot and humid atmosphere (environmental room) | The 1st Time Trial will be performed the week preceding the program training. The 2nd Time Trial will be performed the week following the program training
  The participant has to perform the longer distance possible in 30 min on a stationary bike in hot and humid atmosphere (environmental room). The change of distance (measured in meter) will be assessed before and after the 2 weeks training program.

SECONDARY OUTCOMES:
Change in VO2 Max (ml/kg/min) between pre and post training tests in normal environment | The 1st maximal cardiorespiratory test will be performed the week preceding the program training. The 2nd maximal cardiorespiratory test will be performed the week following the program training
  The participant has to perform a maximal cardiorespiratory test on a stationary bike in normal environment. The change in VO2 Max (measured in ml/kg/min) will be assessed before and after the 2 weeks training program.
Change in Maximal Aerobic Power (Watts) between pre and post training tests in normal environment | The 1st maximal cardiorespiratory test will be performed the week preceding the program training. The 2nd maximal cardiorespiratory test will be performed the week following the program training
  The participant has to perform a maximal cardiorespiratory test on a stationary bike in normal environment. The change in Maximal Aerobic Power (measured in Watts) will be assessed before and after the 2 weeks training program.
Change of "global longitudinal strain of left ventricule" (%) measured during an echocardiography between pre and post training tests in normal environment | The 1st echocardiography will be performed the week preceding the program training. The 2nd echocardiography will be performed the week following the program training
  The participant has to pass an echocardiography with specific measurment of "global longitudinal strain of left ventricule" (united in %). The change will be assessed before and after the 2 weeks training program.
Change on central temperature (°C) between pre and post training test in hot and humid atmosphere (environmental room) | The 1st Time Trial will be performed the week preceding the program training. The 2nd Time Trial will be performed the week following the program training
  Central temperature will be measured during Time Trial in hot and humid atmosphere (environmental room). The change on central temperature (measured in °C) will be assessed before and after the 2 weeks training program.
Change on cutaneours temperature (°C) between pre and post training test in hot and humid atmosphere (environmental room) | The 1st Time Trial will be performed the week preceding the program training. The 2nd Time Trial will be performed the week following the program training
  Cutaneous temperature will be measured during Time Trial in hot and humid atmosphere (environmental room). The change on cutaneours temperature (measured in °C) will be assessed before and after the 2 weeks training program.
Change of Na concentration (mmol/L) in the sweat between pre and post training test in hot and humid atmosphere (environmental room) | The 1st Time Trial will be performed the week preceding the program training. The 2nd Time Trial will be performed the week following the program training
  Sweat quality will be measured during Time Trial in hot and humid atmosphere (environmental room). The change of Na concentration (measured in mmol/l) will be assessed before and after the 2 weeks training program.
Change of body weight loss (Kg) between pre and post training test in hot and humid atmosphere (environmental room) | The 1st measure of body weight will be performed the week preceding the program training. The 2nd measure of body weight will be performed the week following the program training
  Body weight loss will be measured before and after Time Trial in hot and humid atmosphere (environmental room). The change of the body weight (measured in Kg) will be assessed between before and after the 2 weeks training program.
Change of Sleep quality between the first and the last training session of water biking | The sleep self-questionnaire will be performed immediately after the first training session (Day 1) and immediately after the last training session (Day 10) of water biking
  Sleep quality will be measured after the first and the last training session using a specific sleep self-questionnaire (PSQI) to detect the effect of hot or neutral water training during the 2 weeks training program.
  PSQI : Pittsburgh Sleep Quality Index. Qualitative questionnaire, no score measured.
Change of force/velocity power (N/m) between pre and post training test | The 1st measure of force/velocity power will be performed the week preceding the program training. The 2nd measure of force/velocity power will be performed the week following the program training
  The participant has to perform a maximal force/velocity test to measure the force/velocity power on a specific fitness testing cycle (Monark 818 E). The change of force/velocity power (measured in N/m) will be assessed between before and after the 2 weeks training program.
Change of sytemic low grade inflammation (CRP = C-Reactive Protein, mg/l) between pre and post training test | The 1st measure of CRP will be performed the week preceding the program training. The 2nd measure of CRP will be performed the week following the program training
  A blood test will be performed to measure the change of CRP concentration (measured in mg/l) between before and after the 2 weeks training program.
Change of haematocrit (%) between pre and post training test | The 1st measure of haematocrit will be performed the week preceding the program training. The 2nd measure of haematocrit will be performed the week following the program training
  A blood test with complete blood count will be performed to measure the change of haematocrit (which is expressed in %) between before and after the 2 weeks training program.
Change of hemoglobin level (g/100ml) between pre and post training test | The 1st measure of hemoglobin level will be performed the week preceding the program training. The 2nd measure of hemoglobin level will be performed the week following the program training
  A blood test with complete blood count will be performed to measure the change of hemoglobin level (measured in g/100ml) between before and after the 2 weeks training program.
Change of Rate of Perceived Effort (RPE) on a Time Trial between pre and post training tests | The 1st Time Trial will be performed the week preceding the program training. The 2nd Time Trial will be performed the week following the program training
  The Borg Rating of Perceived Exertion (RPE) will be used to measure physical activity intensity level. The scale is from 6 to 20. The higher the score is, the higher the perception of effort is.
  RPE will be measured after the first Time Trial and after the second Time Trial (post training protocol).

CONTACTS AND LOCATIONS:
Locations (1):
- Département de Médecine Physique et Réadaptation, Montpellier, France

REFERENCES:
- [Background] Periard JD, Travers GJS, Racinais S, Sawka MN. Cardiovascular adaptations supporting human exercise-heat acclimation. Auton Neurosci. 2016 Apr;196:52-62. doi: 10.1016/j.autneu.2016.02.002. Epub 2016 Feb 12. PMID 26905458
- [Background] Kelly M, Gastin PB, Dwyer DB, Sostaric S, Snow RJ. Short Duration Heat Acclimation in Australian Football Players. J Sports Sci Med. 2016 Feb 23;15(1):118-25. eCollection 2016 Mar. PMID 26957934
- [Background] Zurawlew MJ, Walsh NP, Fortes MB, Potter C. Post-exercise hot water immersion induces heat acclimation and improves endurance exercise performance in the heat. Scand J Med Sci Sports. 2016 Jul;26(7):745-54. doi: 10.1111/sms.12638. Epub 2015 Dec 9. PMID 26661992
- [Background] Zurawlew MJ, Mee JA, Walsh NP. Post-exercise Hot Water Immersion Elicits Heat Acclimation Adaptations in Endurance Trained and Recreationally Active Individuals. Front Physiol. 2018 Dec 18;9:1824. doi: 10.3389/fphys.2018.01824. eCollection 2018. PMID 30618833
- [Background] Racinais S, Alonso JM, Coutts AJ, Flouris AD, Girard O, Gonzalez-Alonso J, Hausswirth C, Jay O, Lee JK, Mitchell N, Nassis GP, Nybo L, Pluim BM, Roelands B, Sawka MN, Wingo J, Periard JD. Consensus recommendations on training and competing in the heat. Br J Sports Med. 2015 Sep;49(18):1164-73. doi: 10.1136/bjsports-2015-094915. Epub 2015 Jun 11. PMID 26069301
- [Background] Zurawlew MJ, Mee JA, Walsh NP. Post-exercise Hot Water Immersion Elicits Heat Acclimation Adaptations That Are Retained for at Least Two Weeks. Front Physiol. 2019 Aug 28;10:1080. doi: 10.3389/fphys.2019.01080. eCollection 2019. PMID 31555140
- [Derived] Helmer G, Laurent M, Rubio J, Duflos C, Hayot M, Myzia J, Hedon C, Gouzi F, Candau R, Racinais S, Julia M. Training in hot water immersion improved exercise performance in hot and humid conditions in recreational athletes - a randomized controlled trial. Eur J Appl Physiol. 2025 Jul 15. doi: 10.1007/s00421-025-05876-1. Online ahead of print. PMID 40663144